CLINICAL TRIAL: NCT02502383
Title: ACTION PAC: Adolescents Committed to Improvement of Nutrition & Physical Activity
Acronym: ACTION PAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Alberta Kong, MD, MPH, Professor, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01HL118734 (NIH)
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Overweight; Obesity
Keywords: Adolescent; Overweight; Obesity; Weight loss; Nutrition; Physical Activity; School-based; Primary care; Motivational Interviewing
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACTION PAC Behavioral Intervention (Experimental): Students attending intervention schools will receive the ACTION PAC intervention and communication of BMI and other health results to parents via a letter.
  Interventions: Behavioral: ACTION PAC; Behavioral: Communication with parents
- Comparison (Active Comparator): Students attending comparison schools will receive communication of BMI and other health results to parents via a letter.
  Interventions: Behavioral: Communication with parents

INTERVENTIONS:
Behavioral: ACTION PAC — School-based health center providers will use motivational interviewing to assist students with adopting strategies for improving nutrition and increasing physical activity. All participants will receive annual BMI and other health results discussion with clinical providers. Adolescents with overweight/obesity will meet with providers for 16 sessions over 2 years.
  Arms: ACTION PAC Behavioral Intervention
Behavioral: Communication with parents — A letter containing BMI and other health results and obesity prevention recommendations will be sent to parent/guardians.

SUMMARY:
Using a previously created weight management program for adolescents, the intervention will be implemented through school-based health centers (SBHC) and will be delivered by SBHC providers trained in Motivational Interviewing. Students at intervention school sites will be compared to students at control school sites. All students will have baseline, 1 year, and 2 year follow-up to assess if students in the intervention school sites will have improved risk factor profile for metabolic syndrome, improved nutrition and increased physical activity when compared with students at control school sites.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in 9th or 10th grade at participating schools

Exclusion Criteria:

* blood pressure in the range of stage 2 hypertension
* previously diagnosed type 1 or type 2 diabetes
* use of corticosteroids, antipsychotics, metformin, antihypertensive medications, and medications used for dyslipidemia
* inability to perform moderate to vigorous physical activity
* not ambulatory
* a score of 20 or more on Eating Attitudes Test (EAT)-26 screening measure
* developmental disorders that affect weight or ability to understand the study procedures or counseling

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 991 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alberta Kong, MD, MPH, Principal Investigator — UNM Health Sciences Center/Dept of Pediatrics
Locations (1):
- Alberta S Kong, MD, MPH, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Vallabhan MK, Kong AS, Jimenez EY, Summers LC, DeBlieck CJ, Feldstein Ewing SW. Training Primary Care Providers in the Use of Motivational Interviewing for Youth Behavior Change. Res Theory Nurs Pract. 2017 Aug 1;31(3):219-232. doi: 10.1891/1541-6577.31.3.219. PMID 28793946
- [Background] Vallabhan MK, Jimenez EY, Nash JL, Gonzales-Pacheco D, Coakley KE, Noe SR, DeBlieck CJ, Summers LC, Feldstein-Ewing SW, Kong AS. Motivational Interviewing to Treat Adolescents With Obesity: A Meta-analysis. Pediatrics. 2018 Nov;142(5):e20180733. doi: 10.1542/peds.2018-0733. Epub 2018 Oct 22. PMID 30348753
- [Background] Euler R, Jimenez EY, Sanders S, Kuhlemeier A, Van Horn ML, Cohen D, Gonzales-Pacheco D, Kong AS. Rural-Urban Differences in Baseline Dietary Intake and Physical Activity Levels of Adolescents. Prev Chronic Dis. 2019 Jan 3;16:E01. doi: 10.5888/pcd16.180200. PMID 30605423
- [Background] Sanders SG, Jimenez EY, Cole NH, Kuhlemeier A, McCauley GL, Van Horn ML, Kong AS. Estimated Physical Activity in Adolescents by Wrist-Worn GENEActiv Accelerometers. J Phys Act Health. 2019 Sep 1;16(9):792-798. doi: 10.1123/jpah.2018-0344. Epub 2019 Jul 17. PMID 31310994
- [Background] Kuhlemeier A, Jaki T, Jimenez EY, Kong AS, Gill H, Chang C, Resnicow K, Wilson DK, Van Horn ML. Individual differences in the effects of the ACTION-PAC intervention: an application of personalized medicine in the prevention and treatment of obesity. J Behav Med. 2022 Apr;45(2):211-226. doi: 10.1007/s10865-021-00274-2. Epub 2022 Jan 15. PMID 35032253
- [Background] Hess JM, Jimenez EY, Ozechowski TJ, McCauley G, Sanders SG, Sedillo D, Vallabhan MK, Kong AS. Teen and caregiver perspectives on success, clinician role, and family involvement in ACTION PAC, a weight management intervention trial. PEC Innov. 2022 Dec;1:100060. doi: 10.1016/j.pecinn.2022.100060. Epub 2022 Jun 24. PMID 36643597

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from February 2014 to November 2015. Participants were recruited during general school registration events, the classes or practices of interested teachers, and lunch time.
Pre-assignment Details: Teens were excluded based on assessments at the baseline visit: blood pressure in the range of stage 2 hypertension or a score of ≥20 on the Eating Attitudes Test.
Units Other Than Participants: Schools
Groups:
- ACTION PAC: School-based health center providers will use motivational interviewing to assist students with adopting strategies for improving nutrition and increasing physical activity. All participants will receive annual BMI and other health results discussion with clinical providers. Adolescents with overweight/obesity will meet with providers for 16 sessions over 2 years. A letter containing BMI results and obesity prevention recommendations will be sent to parent/guardians.
- Comparison: A letter containing BMI results and obesity prevention recommendations will be sent to parent/guardians.
Period: Overall Study
Arm/Group | ACTION PAC | Comparison
Started | 504; 4 Schools | 487; 4 Schools
Midpoint | 410; 4 Schools | 391; 4 Schools
Completed | 343; 4 Schools | 332; 4 Schools
Not Completed | 161; 0 Schools | 155; 0 Schools
Not completed — Lost to Follow-up | 130 | 131
Not completed — Withdrawal by Subject | 31 | 24

BASELINE CHARACTERISTICS:
Groups:
- ACTION PAC: School-based health center providers will use motivational interviewing to assist students with adopting strategies for improving nutrition and increasing physical activity. All participants will receive annual BMI and other health results discussion with clinical providers. Adolescents with overweight/obesity will meet with providers for 16 sessions over 2 years. A letter containing BMI and other health results and obesity prevention recommendations will be sent to parent/guardians.
- Comparison: A letter containing BMI and other health results and obesity prevention recommendations will be sent to parent/guardians.
- Total: Total of all reporting groups
Arm/Group | ACTION PAC | Comparison | Total
Number analyzed (Participants) | 504 | 487 | 991
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.3 (0.7) | 15.4 (0.7) | 15.3 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 268 | 543
  Male | 229 | 219 | 448
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 451 | 404 | 855
  Not Hispanic or Latino | 53 | 83 | 136
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 504 | 487 | 991
Yearly household income [Count of Participants; unit: Participants]
  <$20,000 | 192 | 206 | 398
  $20,000-39,999 | 163 | 126 | 289
  >=$40,000 | 132 | 137 | 269
  Missing | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Number and Proportion of Participants With Baseline BMI <85th Percentile Who Developed Overweight or Obesity by the End of the Study
Description: Number and percentage of students who had a baseline BMI <85th percentile who had a BMI>= 85th percentile (overweight or obese) at endline
Time Frame: Baseline to two years
Population: Students that had a baseline BMI <85th percentile and who had endline data
Measure: Count of Participants; unit: Participants
Groups:
- ACTION PAC: ACTION PAC: Adolescents enrolled in ACTION PAC will meet with SBHC providers. SBHC providers will use Motivational Interviewing to motivate students to adopt strategies for improving nutrition and increasing physical activity. All participants will receive annual BMI results discussion with providers. Overweight/Obese adolescents will meet with providers for 16 sessions over 2 years.
- Comparison: Comparison: Annual BMI results will not be discussed with participants in comparison schools; however, a letter containing BMI results and obesity prevention recommendations will be sent to parent/guardians.
Arm/Group | ACTION PAC | Comparison
Number analyzed (Participants) | 228 | 206
Participants | 22 | 12

2. Primary Outcome: Change in Physical Activity
Description: Change in minutes of moderate-to-vigorous physical activity as measured by accelerometer for participants who had a baseline BMI <85th percentile and endline data
Time Frame: Baseline to two years
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ACTION PAC | Comparison
Number analyzed (Participants) | 200 | 180
minutes | -14.5 (31.3) | -12.9 (30.7)

3. Primary Outcome: Change in Reported Added Sugar Intake
Description: Reported change in added sugar intake as measured by the Block Kids Food Screener-Last Week for Ages 2-17 for students who had a baseline BMI <85th percentile and endline data
Time Frame: Baseline to two years
Measure: Mean (Standard Deviation); unit: teaspoons
Arm/Group | ACTION PAC | Comparison
Number analyzed (Participants) | 227 | 205
teaspoons | -1.9 (7.8) | -0.9 (6.2)

4. Primary Outcome: Change in Reported Fruit, Vegetables, and Legume Intake (Not Including Potatoes)
Description: Change in reported fruit, vegetables, and legume intake (not including potatoes) for students who had a baseline BMI <85th percentile and endline data
Time Frame: Baseline to two years
Measure: Mean (Standard Deviation); unit: cups
Arm/Group | ACTION PAC | Comparison
Number analyzed (Participants) | 227 | 205
cups | -0.41 (1.42) | -0.32 (1.46)

5. Primary Outcome: Change in BMI Z-score
Description: Change in body-mass index (BMI; weight in kilograms divided by the square of the body height in meters) Z-score for students who had a baseline BMI >= 85th percentile (overweight or obese) and endline data. A Z-score of 0 represents the population mean. A Z-score above 2 indicates obesity (BMI >2 standard deviations above the mean) in children and teens. A decline in BMI Z-score would be a positive outcome in this weight management study.
Time Frame: Baseline to two years
Measure: Mean (Standard Deviation); unit: standard deviation units
Arm/Group | ACTION PAC | Comparison
Number analyzed (Participants) | 119 | 131
standard deviation units | 0.018 (0.302) | -0.047 (0.397)

6. Primary Outcome: Change in HOMA-IR
Description: Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR; insulin resistance index) for students who had a baseline BMI >= 85th percentile (overweight or obese) and endline data. HOMA-IR is calculated using the formula: (fasting glucose [mg/dL] x fasting insulin [microU/mL])/405. HOMA-IR values >2 indicate insulin resistance. A decrease in HOMA-IR would be a positive outcome.
Time Frame: Baseline to two years
Measure: Mean (Standard Deviation); unit: index score units
Arm/Group | ACTION PAC | Comparison
Number analyzed (Participants) | 116 | 129
index score units | 0.613 (5.842) | -0.236 (2.976)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | ACTION PAC | Comparison
All-Cause Mortality (participants affected / at risk) | 0/504 | 0/487
Serious Adverse Events (participants affected / at risk) | 0/504 | 0/487
Other Adverse Events (participants affected / at risk) | 19/504 | 15/487
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACTION PAC (N=504) | Comparison (N=487)
Hospitalization (General disorders) | 15 (15) | 14 (14)
Met criteria for eating disorder (anorexia, bulimia) (Psychiatric disorders) | 3 (3) | 0 (0)
Development of hypertension (Cardiac disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT02502383/Prot_SAP_000.pdf